CLINICAL TRIAL: NCT01461031
Title: Effect of Nefopam on Acute Postoperative Pain in Patients Undergoing Orthognathic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Young Eun Moon, Anesthesiology and Pain Medicine, Clinical Assitant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: nefopam-orthognathic
Record Dates: First submitted 2011-10-11; First posted 2011-10-27 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Pain; Orthognathic Surgery
Keywords: pain; orthognathic
MeSH Terms: conditions — Pain | interventions — Nefopam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: nefopam — nefopam infusion for postoperative 24 hours
Drug: normal saline (control) — normal saline infusion for postoperative 24 hours

SUMMARY:
The aim of this study is to determine the analgesic effect of perioperative nefopam on acute pain in patient undergoing orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-60 years
* undergoing elective orthognathic surgery

Exclusion Criteria:

* pregnancy
* psychiatric disease
* hepatobiliary or renal disease
* monoamine oxidase inhibitor-taking patients

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
pain score on the visual analogue scale | after orthognathic surgery (up to postoperative 24 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St.Mary's Hospital, Seoul, Seocho-gu, South Korea

REFERENCES:
- [Derived] Park HJ, Park JU, Yoo W, Moon YE. Analgesic effects of nefopam in patients undergoing bimaxillary osteotomy: A double-blind, randomized, placebo-controlled study. J Craniomaxillofac Surg. 2016 Feb;44(2):210-4. doi: 10.1016/j.jcms.2015.11.012. Epub 2015 Dec 1. PMID 26725583